CLINICAL TRIAL: NCT00335673
Title: Irbesartan in Mild to Moderate Hypertensive Patients
Brief Title: I SAVE - Irbesartan in Mild to Moderate Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRBES_L_00165
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

INTERVENTIONS:
Drug: Irbesartan (Aprovel) — Aprovel (150 & 300mg) & CoAprovel (300/12.5mg hydrochlorothiazide) one tablet a day per os.

SUMMARY:
* To evaluate control rate of Blood Pressure ≤ 140/90 mm Hg in non-diabetic patients, and ≤ 130/80 mm Hg in diabetic patients.
* To determine percentage of patients achieving blood pressure control according to their profile (naïve, switch, patient history, etc…) at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proved mild to moderate hypertension.
* Newly diagnosed "naïve" hypertensive patients (no prior treatment for hypertension)OR
* Patients who were receiving antihypertensive agents (maximum two - one of them is diuretic) and who in the investigator's opinion would benefit more from switching to the study medication. These patients will undergo a wash out period for not less than 7 days prior to enrollment.

Exclusion Criteria:

* Severe hypertension (Systolic Blood Pressure ≥ 180 mm Hg or Diastolic Blood Pressure ≥ 110 mm Hg).
* Patients with secondary hypertension (for another cause other than type 2 diabetes mellitus).
* Patients with HbA1c > 10%.
* Significant chronic renal impairment (Serum creatinine > 2.0 mg/dL).
* Significant liver disease as shown by SGPT/SGOT (ALAT/ASAT) > 2.5 times the upper limit of the normal range.
* Currently pregnant or lactating females.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Any patient who is in need for a combination antihypertensive therapy from the start (from the medical point of view of his physician).
* Known hypersensitivity to irbesartan, other ARBs (Angiotensin Receptor Blockers), hydrochlorothiazide, or other thiazide diuretics.
* Patients with malignancy during the past 5 years, known collagen disease or severe cardiac, cerebrovascular or gastric disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1630 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Reduction in blood pressure to target values according to ESC 2003 guidelines at the end of the study. | During the study conduct

SECONDARY OUTCOMES:
Occurrence of any side effects leading to treatment discontinuation. | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Mosaad I Morsi, MBBCh, MSc, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Cairo, Egypt